CLINICAL TRIAL: NCT01109719
Title: The Association of ICU Organization and Structure on in Patient Mortality
Brief Title: Critical Illness Outcomes Study
Acronym: CIOS
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Jonathan Sevransky, MD, MHS, Johns Hopkins University
Other Study IDs: CIITG-2; K23GM071399 (NIH)
Record Dates: First submitted 2010-04-22; First posted 2010-04-23 (Estimated); Last update posted 2010-08-25 (Estimated); Status verified 2010-08

CONDITIONS: Critical Illness; Intensive Care; Intensive Care Unit
Keywords: Protocol; Critical pathway; Intensive care units
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
We will test whether the way that an intensive care unit is organized can influence patient related outcomes such as mortality. We will test whether who works in the ICU, and how the ICU is managed will affect the care received by patients. The primary study hypothesis is whether the number of clinical protocols present in an intensive care unit is linked to patient mortality

DETAILED DESCRIPTION:
Title: Do ICU Structural and Procedural Factors Influence Patient Related Outcomes: The Critical Illness Outcome Study (CIOS)

Objectives: This is an exploratory ecologic study designed to examine the organizational and structural factors present in adult intensive care units in the United States. A second objective is to determine whether these organizational and structural factors are associated with patient related outcomes. In addition, we intend to examine whether these organizational and structural issues are associated with patient treatments.

Hypotheses: (Ho) A. The number of protocols used in an ICU is inversely associated with ICU and hospital survival for critically ill patients.

B. Compliance with disease specific protocols is not independently associated with hospital survival for critically ill patients

Specific Aims

1. To describe the organizational structure of participating intensive care units
2. To determine whether the number of protocols used in an intensive care unit is associated with ICU and hospital survival for critically ill patients
3. To determine the frequency with which ICU's follow disease specific protocols for patients with sepsis and ALI

Study Design

1. Prospective ecologic study of 50-60 adult intensive care units and admitted patients
2. ICU organizational and structural data will be collected for each participating ICU
3. 125-200 adult patients in each intensive care unit will be enrolled. Patients within the ICU on a varying, specific day each week will be included. Demographic and treatment variables will be collected for that day on that patient. Outcome data will be collected on ICU and hospital discharge.

ELIGIBILITY:
Inclusion Criteria:

- Hospitalized adult patient in a study ICU on the date of data collection. This includes patients who may be in ICU despite not having critical illness for reasons such as lack of floor beds.

Exclusion Criteria:

-

1. Patient enrolled on previous study collection day 2 Previous enrollment into other study ICU 3. Age < 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients present in study ICU's on the days of enrollement
Sampling Method: Non-Probability Sample
Enrollment: 6000 (Estimated)
Dates: Start 2010-07; Primary Completion 2011-02 (Estimated); Study Completion 2011-04 (Estimated)

PRIMARY OUTCOMES:
In Patient Mortality | Hospital discharge or 60 days

SECONDARY OUTCOMES:
2. Mortality prior to ICU discharge 3. Length of ICU stay 4. Length of hospital stay ICU mortality | ICU discharge or 60 days
ICU length of stay | ICU discharge or 60 days
Length of hospital stay | Hospital discharge or 60 days

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Sevransky, MD, MHS, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Bayview Medical Center, Baltimore, Maryland, United States

REFERENCES:
- [Background] Umoh NJ, Fan E, Mendez-Tellez PA, Sevransky JE, Dennison CR, Shanholtz C, Pronovost PJ, Needham DM. Patient and intensive care unit organizational factors associated with low tidal volume ventilation in acute lung injury. Crit Care Med. 2008 May;36(5):1463-8. doi: 10.1097/CCM.0b013e31816fc3d0. PMID 18434907
- [Background] Levy MM, Rapoport J, Lemeshow S, Chalfin DB, Phillips G, Danis M. Association between critical care physician management and patient mortality in the intensive care unit. Ann Intern Med. 2008 Jun 3;148(11):801-9. doi: 10.7326/0003-4819-148-11-200806030-00002. PMID 18519926
- [Background] Pronovost PJ, Angus DC, Dorman T, Robinson KA, Dremsizov TT, Young TL. Physician staffing patterns and clinical outcomes in critically ill patients: a systematic review. JAMA. 2002 Nov 6;288(17):2151-62. doi: 10.1001/jama.288.17.2151. PMID 12413375
- [Background] Pronovost P, Needham D, Berenholtz S, Sinopoli D, Chu H, Cosgrove S, Sexton B, Hyzy R, Welsh R, Roth G, Bander J, Kepros J, Goeschel C. An intervention to decrease catheter-related bloodstream infections in the ICU. N Engl J Med. 2006 Dec 28;355(26):2725-32. doi: 10.1056/NEJMoa061115. PMID 17192537
- [Derived] Ali NA, Gutteridge D, Shahul S, Checkley W, Sevransky J, Martin GS. Critical Illness Outcome Study: An Observational Study on Protocols and Mortality in Intensive Care Units. Open Access J Clin Trials. 2011 Sep 23;2011(3):55-65. doi: 10.2147/OAJCT.S24223. PMID 25429244